CLINICAL TRIAL: NCT05569291
Title: Investigating the Feasibility of a Physical Activity (tele)coachingv Intervention in Patients with Non-small Cell Lung Cancer: an Explorative Study
Brief Title: Investigating the Feasibility of a Physical Activity (tele)coaching Intervention in Patients with Non-small Cell Lung Cancer: an Explorative Study
Acronym: LUCA-coach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: University Ghent (Other); Jessa Hospital (Other); University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Chris Burtin, Associate Professor, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/160
Record Dates: First submitted 2022-09-16; First posted 2022-10-06 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Non-small Cell Lung Cancer; Non-small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Automated Coaching Program (ACP) (Experimental): The ACP will use the application as developed for patients with COPD and tested to be effective in this population (Demeyer et al., 2017). The program includes 1) one-to-one semi-structured interview (V1) with the coach discussing the importance of physical activity, motivation, self-efficacy, barriers, favorite activities and (coping) strategies to become more active resulting in an individual action plan; 2) step counter (Fitbit; wrist or waist worn) providing direct feedback which automatically sends data to the smartphone via blue-tooth. Patients will be asked to wear this step counter every day during the intervention; 3) smartphone coaching application, installed on a smartphone and linked to the step counter, will provide automated coaching by displaying an individual activity goal (expressed as daily step count) and daily and weekly feedback on the performance (steps) of the patient. 4) phone calls by the coaches initiated in pre-defined situations.
  Interventions: Device: Automated Coaching Program (ACP)
- Manual Coaching Program (MCP) (Experimental): The MCP includes 1) one-to-one semi-structured interview (V1) with the coach discussing the importance of physical activity, motivation, self-efficacy, barriers, favorite activities and (coping) strategies to become more active resulting in an individual action plan; 2) step counter (Fitbit, wrist or waist worn), that will be linked with a smartphone using the Fitbit application providing direct feedback. Patients can access the Fitbit application if they want to, but they will not receive personal feedback; 3) weekly phone calls by the coaches, interviewing patients on their progress, performance (steps) and feedback. The first goal is based on the physical activity level at the beginning of the coaching intervention (median of 4 days). The individual activity goal (expressed as daily step count) will be revised based on the patient's willingness to increase.
  Interventions: Other: Manual Coaching Program (MCP)

INTERVENTIONS:
Device: Automated Coaching Program (ACP) — A semiautomated tele coaching program (application installed on a smartphone device with real time feedback and motivational messages) and a step counter (Fitbit Charge 4) providing direct feedback on total daily number of steps, walking time, time in at least moderate PA and movement intensity during walking.
  Arms: Automated Coaching Program (ACP)
Other: Manual Coaching Program (MCP) — A telecoaching program using a step counter (Fitbit Charge 4) without this custom smartphone application but with the Fitbit application. This intervention will be more focused on weekly personal feedback from a coach by telephone.
  Arms: Manual Coaching Program (MCP)

SUMMARY:
The aim of this study is to investigate the acceptability, actual usage, feasibility and safety of 1) a (semi) automated PA tele coaching intervention including smartphone application and stepcounter (Fitbit Charge 4) and 2) a manual PA tele coaching program using only a stepcounter (Fitbit Charge 4) without custom smartphone application but still linked with a smartphone using the Fitbit application and to make population specific adaptations to the intervention for patients with NSCLC after lung resection surgery.

ELIGIBILITY:
Inclusion Criteria:

* Three to nine months after a lung resection surgery for non-small cell lung cancer
* If patients received adjuvant chemotherapy, the inclusion window will be three months to nine months after the end of adjuvant chemotherapy
* Adults (+18 year)

Exclusion Criteria:

* Progressive or recurrent lung cancer
* Who had other malignancies in the last 2 years
* Psychiatric disorders
* Other ongoing treatments
* Involved in or planned to start a multidisciplinary rehabilitation program
* Unable to learn to work with a new electronic device (e.g. smartphone)
* Not understanding and speaking Dutch
* Patients with comorbidities precluding them from participation in a physical activity intervention

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of the coaching programs | 9 weeks after the inclusion of the patient
  (i.e. to what extent patients receiving the intervention consider it as appropriate) Acceptability will be assessed through quantitative data (a project-tailored questionnaire) and qualitative data collection (patient interview with open questions).
  Patients will be asked to fill in a self-administered, project-tailored, multiple choice questionnaire on their experiences with the intervention.
  Patient interviews with open questions will be conducted by the local PA coach in each center.
Actual usage of the coaching programs | During the whole 8-week intervention
  (i.e. the degree to which patients use the components of the intervention as it was designed) Actual usage of the custom application by patients will be assessed objectively through the smartphone app log (for participants in the ACP group). This will include information about completion of the app tasks and step counter data on a day-by-day basis and will be automatically collected in the back-end of the application.
  Actual usage of the step counter (for participants in both intervention groups) will be defined based on the presence of step count data (ie, ≥70 steps for that day). The frequency at which patients looked at their step counter will be assessed subjectively in the project-tailored questionnaire.
Feasibility of the coaching programs | 9 weeks after the inclusion of the patient
  (i.e. the extent to which the treatment can be successfully used within a given setting). Feasibility will be assessed through quantitative data (a project-tailored questionnaire) and qualitative data collection (patient interview with open questions).
  Patients will be asked to report the smartphone intervention and use of the step counter and indicate if it was not too much of a burden to work with when they are asked how they have experienced the technical aspects of the intervention. Coaches will collect contact time with patients and preparation time in a logbook in an Excel file. Also, how many times patients are contacted and the number of technical problems will be collected.
Safety of the coaching programs | During the whole 8-week intervention
  Detailed information of any adverse event (AE) will be collected during the pilot phase. Description, severity, start and stop, seriousness, outcome and relation to the intervention will be described for every reported AE. If problems occur during the intervention, patients are asked to contact the coach to discuss possible AE's. If necessary, an extra visit or consultation with a physician will be scheduled. During each patient contact coaches will also seek information on AE's. All events, whether reported by the patient or noted by the coach, will be recorded in the patient's medical record and in the (e)CRF within a reasonable time after becoming aware.

SECONDARY OUTCOMES:
Physical activity | 1 whole week after inclusion and 1 whole week after the 8-week intervention
  PA will be objectively measured using the Dynaport Movemonitor (DAM, McRoberts, The Hague, The Netherlands), a small (106.6 x 58 x 11.5mm), light-weight CE marked tri-axial accelerometer with a sampling frequency of 100Hz. The Dynaport Movemonitor analyzes and expresses digital data not only in terms of locomotion and movement parameters, but also in terms of body posture. Data will be processed with commercially available software (MoveMonitor; McRoberts B.V., The Hague, The Netherlands). The monitor will be worn at the waist level using a comfortable elastic strap.
  Patients will wear the monitor during 1 week before and after the intervention. They will be asked to wear the device continuously, except during bathing/showering and sleeping. Days with less than 8 hours of wearing time will be excluded from the analysis. Patients will not be included in the analysis if they did not have at least 4 valid weekdays of measurement.
Functional exercise capacity | 1 week before the start of the intervention and immediately after the 8-week intervention
  Functional exercise capacity will be measured using a six-minute walk distance (6MWD) test. This test is a routinely used, valid, reliable and safe exercise test in patients with chronic respiratory diseases. The test is standardized in a 30m corridor and will be performed according to the protocol proposed by ERS/ATS.
  Heart rate and oxygen saturation are measured before, during and after the test. Symptom scores for dyspnea and leg fatigue are assessed, at the beginning and end of the test, by the BORG scale. The 6MWD will be measured twice per visit.
Symptoms | 1 week before the start of the intervention and immediately after the 8-week intervention
  The modified medical research council (MMRC) dyspnea scale is a simple one- question grading system to assess the patient's symptoms of breathlessness in daily life. The Multidimensional Fatigue Inventory (MFI-20) is a 20-item self-report instrument designed to measure fatigue, a cardinal symptom in cancer survivors. It covers the following dimensions: general fatigue, physical fatigue, reduced activity, reduced motivation and mental fatigue.
Quality of Life - EORTC QLQ-C30-LC13 | 1 week before the start of the intervention and immediately after the 8-week intervention
  The European Organization for the Research and Treatment of Cancer Questionnaire and lung cancer module (EORTC QLQ-C30-LC13) is a clinically valid and useful tool for assessing disease- and treatment-specific symptoms in lung cancer patients participating in clinical trials, when combined with the EORTC core quality of life questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Burtin, PhD, Principal Investigator — University Hasselt; Heleen Demeyer, PhD, Principal Investigator — University Ghent
Locations (2):
- Belgium (2):
  - REVAL Gebouw A, Diepenbeek, Limburg
  - UZ Gent, Ghent, Oost-Vlaanderen

IPD SHARING:
Plan to Share IPD: No